CLINICAL TRIAL: NCT04222712
Title: A Randomized, Double-Masked, Dose-Ranging Study to Evaluate the Safety and Tolerability of TRS01 Eye Drops in Participants With Active Non-infectious Anterior Uveitis.
Brief Title: A Study to Evaluate TRS01 Eye Drops in Participants With Active Non-infectious Anterior Uveitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tarsier Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GADOT 20/20
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-08

CONDITIONS: Non-infectious Anterior Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRS01 low dose (Experimental)
  Interventions: Drug: TRS01 eye drops
- TRS01 high dose (Experimental)
  Interventions: Drug: TRS01 eye drops

INTERVENTIONS:
Drug: TRS01 eye drops — Dosed four times a day (QID)
  Arms: TRS01 low dose
Drug: TRS01 eye drops — Dosed four times a day (QID)
  Arms: TRS01 high dose

SUMMARY:
The objective of this study is to evaluate the safety of TRS01 eye drops in participants with active non-infectious anterior uveitis

.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to provide informed consent, follow instructions and complete all required study visits for the duration of the study.
* Diagnosed with active non-infectious anterior uveitis requiring an increase or initiation of topical steroids for management of ocular inflammation.

An eligible subject must have:

* Non-infectious active anterior uveitis with anterior chamber cells Grade 2 or Grade 3, as specified per protocol.
* Must have vision ≥ 20/40 in the non-study eye.
* Use adequate birth control by men and women, if of reproductive potential and sexually active, as specified per protocol.

Exclusion Criteria:

* Any form of infectious uveitis
* Active retinitis
* Cancer or melanoma that is actively treated with immunotherapy
* Pregnancy / lactation
* Receiving specific medication/interventions as specified per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Palisades Park, Palisades Park, New Jersey
  - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRS01 Low Dose | TRS01 High Dose
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRS01 Low Dose | TRS01 High Dose | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (13.44) | 56.0 (12.45) | 52.6 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Iris color [Count of Participants; unit: Participants]
  Dark brown | 4 | 2 | 6
  Light brown | 0 | 3 | 3
  Blue | 0 | 1 | 1
  Green | 1 | 1 | 2
  Hazel | 3 | 1 | 4
Anterior Chamber Cell Grade in the study eye [Count of Participants; unit: Participants] — A scale of 0 to 4, where Grade 0 = No ACC and Grade 4 = Severe ACC level. i.e., higher scores are considered worse outcomes
  Participants
    2 | 6 | 2 | 8
    3 | 2 | 6 | 8
Disease course [Count of Participants; unit: Participants]
  Acute | 3 | 2 | 5
  Acute on Chronic | 4 | 3 | 7
  Chronic | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Both Systemic and Ocular Adverse Events
Description: Number of patients experiencing Adverse Events during the study
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TRS01 Low Dose | TRS01 High Dose
Number analyzed (Participants) | 8 | 8
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | TRS01 Low Dose | TRS01 High Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRS01 Low Dose (N=8) | TRS01 High Dose (N=8)
Anxiety (Psychiatric disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 — Judged by PI to be unrelated to study drug
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Instillation site pain (General disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Fatigue (General disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Nausea (Gastrointestinal disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Iritis (Eye disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Diarrhoea (Gastrointestinal disorders) | 1 | 0 — Judged by PI to be unrelated to study drug
Headache (Nervous system disorders) | 1 | 0 — Judged by PI to be unrelated to study drug
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 — Judged by PI to be unrelated to study drug
Hordeolum (Infections and infestations) | 1 | 0 — Judged by PI to be unrelated to study drug
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Syphilis (Infections and infestations) | 0 | 1 — Judged by PI to be unrelated to study drug
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 — Judged by PI to be unrelated to study drug
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 — Judged by PI to be unrelated to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT04222712/Prot_SAP_000.pdf